CLINICAL TRIAL: NCT00537316
Title: Comparison of the Efficacy and Safety of Infliximab, as Monotherapy or in Combination With Azathioprine, Versus Azathioprine Monotherapy in Moderate to Severe Active Ulcerative Colitis (Part 1) Comparison of Maintenance Versus Intermittent Infliximab Treatment in Maintaining Remission: A Follow-Up of Efficacy and Safety (Part 2)
Brief Title: Efficacy & Safety of Infliximab Monotherapy Vs Combination Therapy Vs AZA Monotherapy in Ulcerative Colitis (Part 1) Maintenance Vs Intermittent Therapy for Maintaining Remission (Part 2)(Study P04807)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Infusion reactions during re-induction cycles after a period of no treatment in another study [P04563, NCT0358670]
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04807
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Infliximab (IFX) (Experimental): Part 1: IFX 5 mg/kg of body weight intravenous (IV) infusions was to be administered at Weeks 0, 2, and 6 and placebo to AZA was to be taken orally every day for 16 weeks. Responders to IFX at Week 8, were to receive one more IFX infusion at Week 14; non-responders to IFX were to receive placebo IFX infusions at Weeks 8 and 10 and an additional IFX infusion at Week 14. Part 2: Participants in steroid-free remission at Week 16 of Part 1 were to be randomized to either maintenance (every 8 weeks [q8w]) or intermittent (upon relapse) open-label IFX (last IFX infusion administered at Week 86) plus double-blind oral AZA/placebo treatment as allocated in Part 1 (last dose at the final visit, Week 94). Responders at Week 16 who had not achieved steroid-free remission were to continue to receive IFX infusions every 8 weeks.
  Interventions: Biological: Infliximab (IFX); Drug: Placebo to Azathioprine; Drug: Placebo infusion
- Azathioprine (AZA) (Active Comparator): AZA 2.5 mg/kg of body weight orally every day for 16 weeks. Responders to AZA monotherapy at Week 8 were to continue on AZA therapy and receive one placebo infusion at Week 14; non-responders to AZA at Week 8 would be eligible to receive an IFX infusion at Weeks 8, 10, and 14. Participants in steroid-free remission at Week 16 were to continue on AZA monotherapy and were to be followed up for safety in Part 2. Participants who experienced a relapse of disease after Week 16 were to continue daily AZA monotherapy and receive 3 infusions of IFX (induction therapy at Weeks 0, 2, and 6) followed by infusions every 8 weeks (maintenance therapy).
  Interventions: Drug: Azathioprine (AZA); Drug: Placebo infusion
- IFX/AZA (Experimental): IFX 5 mg/kg of body weight IV infusions at Weeks 0, 2, and 6 plus AZA 2.5 mg/kg orally every day for 16 weeks. Responders to IFX/AZA at Week 8 were to receive one more IFX infusion at Week 14; non-responders to IFX/AZA were to receive placebo infusions at Weeks 8 and 10 and one additional IFX infusion at Week 14. Part 2: Participants in steroid-free remission at Week 16 of Part 1 were to be randomized to either maintenance (every 8 weeks [q8w]) or intermittent (upon relapse) open-label IFX (last IFX infusion administered at Week 86) plus double-blind oral AZA/placebo treatment as allocated in Part 1 (last dose at the final visit, Week 94). Responders at Week 16 who had not achieved steroid-free remission were to continue to receive IFX infusions every 8 weeks.
  Interventions: Biological: Infliximab (IFX); Drug: Azathioprine (AZA); Drug: Placebo infusion
- Maintenance IFX/AZA (during Part 2) (Experimental): Participants randomized to maintenance IFX/AZA in Part 2 of the study were to receive IFX 5 mg/kg of body weight IV infusions every 8 weeks (beginning at Week 22, Week 6 for direct entry) plus AZA 2.5 mg/kg of body weight daily. Four participants were from Part 1 of the study and 1 participant was enrolled directly into Part 2 of the study.
  Interventions: Biological: Infliximab (IFX); Drug: Azathioprine (AZA)
- Maintenance IFX (during Part 2) (Experimental): Participants randomized to maintenance IFX were to receive IFX 5 mg/kg of body weight IV infusions every 8 weeks (beginning at Week 22, Week 6 for direct entry) in Part 2 of the study. Placebo to AZA therapy was to continue as allocated in Part 1 of the study. All participants were from Part 1 of the study.
  Interventions: Biological: Infliximab (IFX)
- Intermittent IFX/AZA (during Part 2) (Experimental): Participants randomized to intermittent IFX/AZA were to receive IFX 5 mg/kg of body weight IV infusions only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained) plus AZA 2.5 mg/kg of body weight daily in Part 2 of the study. Three participants were from Part 1 of the study and 1 participant was enrolled directly into Part 2 of the study.
  Interventions: Biological: Infliximab (IFX); Drug: Azathioprine (AZA)
- Intermittent IFX (during Part 2) (Experimental): Participants randomized to intermittent IFX were to receive IFX 5 mg/kg of body weight IV infusions only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained). Placebo to AZA therapy was to continue as allocated in Part 1 of the study. One participant was from Part 1 of the study and 1 participant was enrolled directly into Part 2 of the study.
  Interventions: Biological: Infliximab (IFX)

INTERVENTIONS:
Biological: Infliximab (IFX) — IFX intravenous (IV) infusion dosed at 5mg/kg of body weight
  Other Names: Remicade
  Arms: IFX/AZA; Infliximab (IFX); Intermittent IFX (during Part 2); Intermittent IFX/AZA (during Part 2); Maintenance IFX (during Part 2); Maintenance IFX/AZA (during Part 2)
Drug: Azathioprine (AZA) — AZA 50 mg tablet dosed at 2.5 mg/kg of body weight orally every day
  Other Names: Imuran
  Arms: Azathioprine (AZA); IFX/AZA; Intermittent IFX/AZA (during Part 2); Maintenance IFX/AZA (during Part 2)
Drug: Placebo to Azathioprine — Placebo to AZA tablet orally every day
  Arms: Infliximab (IFX)
Drug: Placebo infusion — Placebo to IFX intravenous (IV) infusion
  Arms: Azathioprine (AZA); IFX/AZA; Infliximab (IFX)

SUMMARY:
Part 1 of this study is a 3-arm, randomized, active-controlled, parallel-group, multicenter, double-blind, double-dummy, 16-week study to compare the efficacy and safety of infliximab (IFX), as monotherapy or in combination with azathioprine (AZA) versus AZA monotherapy in adults with moderate to severe active ulcerative colitis (UC). Participants who qualify at the Baseline Visit will be eligible to be randomized to one of the three active treatment groups.

Participants in the IFX/AZA combination therapy and IFX monotherapy cohorts will receive IFX infusions at Weeks 0, 2, and 6 and daily oral AZA/placebo, respectively; participants in the AZA cohort will receive daily oral AZA and placebo infusions at Weeks 0, 2, and 6. At Week 8, all participants will be evaluated for response.

Participants responding to IFX treatment at Week 8, either as monotherapy or in combination with AZA, will receive one more IFX infusion at Week 14; non-responders to IFX therapy will receive placebo infusions at Weeks 8 and 10 and one additional IFX infusion at Week 14.

Participants responding to AZA monotherapy at Week 8 will continue on AZA therapy and receive one placebo infusion at Week 14; nonresponders to AZA will be eligible to receive IFX at Weeks 8, 10, and 14.

Part 2: Participants in remission on IFX monotherapy or IFX/AZA treatment at Week 16 will be randomized to either maintenance or intermittent open-label IFX treatment; randomization will be stratified based on oral AZA/placebo treatment in Part 1. Oral AZA/placebo treatment will continue to be double-blinded. All participants will continue to receive oral AZA/ placebo for the duration of the study.

Participants randomized to maintenance IFX treatment will receive scheduled IFX infusions every 8 weeks beginning at Week 22 (Week 6 for direct entry). If participants lose response, or if treatment has to be discontinued because of an adverse event, these participants are considered treatment failures, and should be followed up for safety at the scheduled 6-month visits (Weeks 38, 62, and 94 [Weeks 22, 46, and 78 for direct entry]). These participants will receive standard of care per their personal physician.

Participants randomized to intermittent IFX treatment will be evaluated every 8 weeks. Participants will receive IFX only upon relapse of disease. Treatment with IFX will be initiated at Weeks 0, 2, and 6 of the individual treatment cycle and will continue every 8 weeks until remission is regained. Throughout the study, individual treatment cycles will be repeated whenever a subject relapses.

In addition, to facilitate enrollment into Part 2, participants who received treatment outside of Part 1 and who are in remission on IFX with or without AZA/6-mercaptopurine (6-MP) will be allowed to enter directly into Part 2. In the Czech Republic, direct entry into Part 2 of the study is not allowed.

A higher than expected incidence of serious infusion reactions observed in the intermittent treatment arm of another study (Protocol P04563, NCT0358670) conducted in participants with moderate to severe psoriasis resulted in the termination of that study. Based on the similarities in study design between the intermittent treatment arm of P04563 and the intermittent treatment arm of Part 2 of this study, enrollment to Part 2 of this study was put on hold, for precautionary reasons. At the same time, all participants already enrolled in the intermittent treatment arm of Part 2 were asked to discontinue from the trial. In October 2009, a decision was made by the sponsor to terminate the whole study (Part 1 and 2). At that time, participants enrolled in Part 1 of the study were allowed to complete their treatment up to Week 16.

ELIGIBILITY:
Inclusion Criteria:

* must be >=21 years of age at the time of informed consent, of either sex, and of any race;
* must have endoscopic evidence of UC, as determined by sigmoidoscopy, within 14 days prior to Baseline;
* must have a total Mayo score of 6 to 12 points at Baseline;
* must have responded inadequately to corticosteroid treatment (ie, the last or current UC flare did not respond adequately to a standard course of corticosteroids) with or without 5 aminosalicylic acid (5-ASA);
* must be off corticosteroids or on a stable dose of corticosteroid for at least 2 weeks prior to enrollment. The maximal daily dose of corticosteroid at Baseline must not exceed the equivalent of 30 mg of prednisone;
* must be naïve to infliximab and other tumor necrosis factor-alpha (TNF-α) antagonists;
* must be either naïve to AZA/6-MP or have not received AZA/6-MP for at least 3 months before enrollment in the study;
* considered eligible according to the following tuberculosis (TB) screening criteria:

  * have no history of latent or active TB prior to Screening;
  * have no signs or symptoms suggestive of active TB upon medical history and/or physical examination;
  * have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of IFX;
  * within 1 month prior to the first administration of infliximab, either have negative tuberculin skin test OR have a newly identified positive tuberculin test during Screening in which active TB has been ruled out, and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of IFX.
  * must have a chest X-ray (posterior-anterior and lateral views), taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current active TB or old active TB;
* have had UC for more than 10 years should have had a full colonoscopy within 2 years prior to Screening for the surveillance of dysplasia;
* screening and Baseline clinical laboratory tests (complete blood count [CBC] and blood chemistries) must be within predetermined parameters
* had been on antibiotics for the treatment of UC (eg, ciprofloxacin and metronidazole) must have been discontinued from them at least 3 weeks prior to Screening;
* must be free of any clinically significant condition or situation, other than UC that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study;
* willing and able to adhere to the study visit schedule and other protocol requirements;
* capable of providing written informed consent, which must be obtained prior to conducting any protocol-specified procedures;
* women of child-bearing potential and all men must agree to use a medically accepted method of contraception prior to screening, while receiving protocol-specified medication, and for 6 months after stopping the medication. Acceptable methods of contraception include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device (IUD), oral or injectable hormonal contraceptive, and surgical sterilization (eg, hysterectomy or tubal ligation). Women of child-bearing potential who are not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study;
* female participants of childbearing potential must have a negative serum pregnancy test (beta-human chorionic gonadotropin) at Screening and a negative urine pregnancy test at Baseline.

Exclusion Criteria:

* have severe extensive colitis as evidenced by:

  * investigator judgment that the participant is likely to require colectomy within 12 weeks of Baseline

OR

* at least 4 of these symptoms at Screening or Baseline visits, as follows:

  * diarrhea with >=6 bowel movements/day with macroscopic blood in stool;
  * focal severe or rebound abdominal tenderness;
  * persistent fever (>=37.5 degrees C) for at least 3 days prior to baseline;
  * tachycardia (>100 beats/minute);
  * hemoglobin <8.5 g/dL (5.3 mM/L).

    * require, or are required within the 2 months prior to baseline, surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage or other conditions possibly confounding the evaluation of disease activity;
    * have severe, fixed symptomatic stenosis of the large or small intestine;
    * have current evidence of colonic obstruction or history within the 6 months prior to baseline, confirmed with objective radiographic or endoscopic evidence of a stricture with resulting obstruction (dilation of the colon proximal to the stricture on barium radiograph or an inability to traverse the stricture at endoscopy);
    * have a history of colonic mucosal dysplasia;
    * presence on screening endoscopy of adenomatous colonic polyps, if not removed prior to study entry, or history of adenomatous colonic polyps that were not removed;
    * have the presence of a stoma;
    * have a history of extensive colonic resection that would prevent adequate evaluation of clinical disease activity (eg, less than 30 cm of colon remaining);
    * have had a positive stool culture for enteric pathogens, pathogenic ova or parasites within 4 months prior to Baseline unless participant has received treatment and had a negative stool examination 1 week or longer after the end of treatment;
    * have a concomitant diagnosis of congestive heart failure (CHF), including medically controlled asymptomatic subjects;
    * have had serious infections (eg, active hepatitis, pneumonia, or pyelonephritis) within 2 months of Screening. Less serious infections (such as acute upper respiratory tract infection [colds] or a simple urinary tract infection) need not be considered as an exclusion at the discretion of the investigator;
    * have had a nontuberculous mycobacterial infection or opportunistic infection (eg, cytomegalovirus, Pneumocystis carinii, aspergillosis) within 6 months prior to Screening;
    * have a known infection with human immunodeficiency virus (HIV) and/or hepatitis B or hepatitis C;
    * have a history of a known allergy to murine proteins or allergy/sensitivity to study drug or its excipients;
    * have current signs and symptoms of systemic lupus erythematosus, or severe, progressive, or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic, or cerebral diseases;
    * have a known history of demyelinating disease suggestive of multiple sclerosis or optic neuritis;
    * presence of a transplanted organ (with the exception of a corneal transplant >3 months prior to Screening);
    * have a history of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (eg, nodes in the posterior triangle of the neck, infra-clavicular, epitrochlear, or periaortic areas), or splenomegaly;
    * have any current known malignancy or malignancy within 5 years prior to Screening (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence);
    * have poor tolerability of venipuncture or lack of adequate venous access for required blood sampling and infusion of study drug during the study period;
    * have had a known substance abuse or dependency (drug or alcohol) within 3 years of Screening;
    * require chronic (>=1 month) and frequent use (>=3 days per week)of nonsteroidal anti-inflammatory drugs (NSAIDs) except low-dose aspirin for prevention of heart attacks, unstable angina, or transient ischemic attacks;
    * have other inflammatory diseases that might interfere with the evaluation of the ulcerative colitis;
    * have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to Screening.
    * have had a Bacille Calmette-Guerin (BCG) vaccination within 12 months of Screening.
    * have had a chest X-ray within the 3 months prior to the first administration of study agent that shows an abnormality suggestive of malignancy or current active infection, including TB.
    * have received any specified prohibited treatment more recently than the indicated washout period prior to Screening;
    * who are participating in any other clinical study or who have received treatment with any investigational drug or device within 3 months prior Screening;
    * who is part of the staff or a family member of the staff personnel directly involved with this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Panaccione R, Ghosh S, Middleton S, Marquez JR, Scott BB, Flint L, van Hoogstraten HJ, Chen AC, Zheng H, Danese S, Rutgeerts P. Combination therapy with infliximab and azathioprine is superior to monotherapy with either agent in ulcerative colitis. Gastroenterology. 2014 Feb;146(2):392-400.e3. doi: 10.1053/j.gastro.2013.10.052. PMID 24512909
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were randomized but not treated. Part 1: 237 participants received ≥1 dose study medication. Part 2: Of 108 enrolled/randomized participants, 95 continued assigned treatment from Part 1 and 13 were randomized and entered into Part 2 of the study (10 participants from Part 1 and 3 participants who were enrolled directly into Part 2).
Groups:
- Infliximab (IFX): IFX 5 mg/kg Intravenous (IV) infusions administered at Weeks 0, 2, and 6 and placebo to AZA (orally) daily for 16 weeks. Responders to IFX at Week 8, will receive one more IFX infusion at Week 14; non-responders to IFX will receive placebo infusions at Weeks 8 and 10 and an additional IFX infusion at Week 14.
- Azathioprine (AZA): AZA 2.5 mg/kg orally for 16 weeks and placebo to IFX infusion at Weeks 0, 2, and 6. Responders to AZA monotherapy at Week 8 will continue on AZA therapy and receive one placebo IFX infusion at Week 14; non-responders to AZA at Week 8 will be eligible to receive IFX at Weeks 8, 10, and 14. This group included 20 participants who did not respond to AZA monotherapy at Week 8 had IFX added to their treatment regimen at Weeks 8, 10, and 14.
- IFX/AZA: IFX 5 mg/kg IV infusion at Weeks 0, 2, and 6 plus AZA 2.5 mg/kg orally daily for 16 weeks.
  Responders to IFX/AZA at Week 8 will receive one more IFX infusion at Week 14; non-responders to IFX/AZA will receive placebo IFX infusions at Weeks 8 and 10 and one additional IFX infusion at Week 14.
- Maintenance IFX/AZA (During Part 2): Participants randomized to maintenance IFX/AZA received IFX 5 mg/kg of body weight every 8 weeks (beginning at Week 22, Week 6 for direct entry) plus AZA 2.5 mg/kg of body weight daily in Part 2 of the study (4 participants from Part 1 of the study and 1 participant was enrolled directly into Part 2 of the study).
- Maintenance IFX (During Part 2): Participants randomized to maintenance IFX received infusion of IFX 5 mg/kg of body weight every 8 weeks (beginning at Week 22, Week 6 for direct entry) and placebo to AZA therapy as allocated in Part 1 of the study (all participants were from Part 1 of the study).
- Intermittent IFX/AZA (During Part 2): Participants randomized to intermittent IFX/AZA received IFX 5 mg/kg of body weight only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained) plus AZA 2.5 mg/kg of body weight daily in Part 2 of the study (3 participants from Part 1 of the study and 1 participant was enrolled directly into Part 2 of the study).
- Intermittent IFX (During Part 2): Participants randomized to intermittent IFX received IFX 5 mg/kg of body weight only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained) and placebo to AZA as allocated in Part 1 of the study (1 participant from Part 1 of the study and 1 participant was enrolled directly into Part 2 of the study).
Period: Part 1
Arm/Group | Infliximab (IFX) | Azathioprine (AZA) | IFX/AZA | Maintenance IFX/AZA (During Part 2) | Maintenance IFX (During Part 2) | Intermittent IFX/AZA (During Part 2) | Intermittent IFX (During Part 2)
Started | 79 | 80 | 80 | 0 | 0 | 0 | 0
Completed | 65 | 53 | 63 | 0 | 0 | 0 | 0
Not Completed | 14 | 27 | 17 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 11 | 8 | 0 | 0 | 0 | 0
Not completed — Protocol defined clinical event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 8 | 4 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 5 | 1 | 0 | 0 | 0 | 0
Not completed — Did not meet protocol eligibility | 1 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Administrative | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Infliximab (IFX) | Azathioprine (AZA) | IFX/AZA | Maintenance IFX/AZA (During Part 2) | Maintenance IFX (During Part 2) | Intermittent IFX/AZA (During Part 2) | Intermittent IFX (During Part 2)
Started | 37 | 10 | 48 | 5 | 2 | 4 | 2
Completed | 11 | 1 | 16 | 2 | 1 | 0 | 0
Not Completed | 26 | 9 | 32 | 3 | 1 | 4 | 2
Not completed — Never entered follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 4 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Administrative | 16 | 8 | 24 | 3 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Infliximab (IFX): All treated participants. IFX 5 mg/kg IV infusions administered at Weeks 0, 2, and 6 and placebo to AZA daily for 16 weeks. Responders to IFX at Week 8, will receive one more IFX infusion at Week 14; non-responders to IFX will receive placebo infusions at Weeks 8 and 10 and an additional IFX infusion at Week 14.
- Azathioprine (AZA): All treated participants. AZA 2.5 mg/kg orally for 16 weeks and placebo to IFX infusion at Weeks 0, 2, and 6. Responders to AZA monotherapy at Week 8 will continue on AZA therapy and receive one infliximab placebo infusion at Week 14; non-responders to AZA at Week 8 will be eligible to receive infliximab at Weeks 8, 10, and 14. This group included 20 participants who did not respond to AZA monotherapy at Week 8 had IFX added to their treatment regimen at Weeks 8, 10, and 14.
- IFX/AZA: All treated participants. IFX 5 mg/kg IV at Weeks 0, 2, and 6 plus AZA 2.5 mg/kg orally daily for 16 weeks.
  Responders to IFX/AZA at Week 8 will receive one more infliximab infusion at Week 14; non-responders to IFX/AZA will receive placebo IFX infusions at Weeks 8 and 10 and one additional IFX infusion at Week 14.
- Maintenance IFX/AZA (During Part 2): Participants enrolled directly and randomized to maintenance IFX/AZA received IFX 5 mg/kg of body weight every 8 weeks (beginning at Week 22, Week 6 for direct entry) plus AZA 2.5 mg/kg of body weight daily in Part 2 of the study (4 participants from Part 1 of the study and 1 participant enrolled directly into Part 2 of the study).
- Intermittent IFX/AZA (During Part 2): Participants enrolled directly and randomized to intermittent IFX/AZA received IFX 5 mg/kg of body weight only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained) plus AZA 2.5 mg/kg of body weight daily in Part 2 of the study (3 participants from Part 1 of the study and 1 participant enrolled directly into Part 2 of the study).
- Intermittent IFX (During Part 2): Participants enrolled directly and randomized to intermittent IFX received IFX 5 mg/kg of body weight only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained) and placebo to AZA daily in Part 2 of the study (1 participant from Part 1 of the study and 1 participant enrolled directly into Part 2 of the study).
- Total: Total of all reporting groups
Arm/Group | Infliximab (IFX) | Azathioprine (AZA) | IFX/AZA | Maintenance IFX/AZA (During Part 2) | Intermittent IFX/AZA (During Part 2) | Intermittent IFX (During Part 2) | Total
Number analyzed (Participants) | 78 | 79 | 80 | 1 | 1 | 1 | 240
Age, Customized [Number; unit: Participants] — Baseline characteristics for Part 2 are presented for the direct entry participants only: 1 participant randomized to the maintenance IFX/AZA group, 1 participant randomized to the intermittent IFX/AZA group, and 1 participant randomized to the intermittent IFX group. No participants were directly enrolled into the maintenance IFX group in Part 2 of the study.
  Participants
    <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
    18 years to <65 years | 77 | 76 | 78 | 1 | 1 | 1 | 234
    65 years and older | 1 | 3 | 2 | 0 | 0 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics for Part 2 are presented for the direct entry participants only: 1 participant randomized to the maintenance IFX/AZA group, 1 participant randomized to the intermittent IFX/AZA group, and 1 participant randomized to the intermittent IFX group. No participants were directly enrolled into the maintenance IFX group in Part 2 of the study.
  Participants
    Female | 36 | 46 | 32 | 0 | 1 | 1 | 116
    Male | 42 | 33 | 48 | 1 | 0 | 0 | 124

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants in Steroid-free Remission at Week 16
Description: Steroid-free remission is defined as a total Mayo score of 2 points or lower, with no individual sub-score exceeding 1 point, without the use of corticosteroids. The total Mayo score consists of the following 4 sub-scores: stool frequency, rectal bleeding, findings of endoscopy (sigmoidoscopy), and physician's global assessment.
Time Frame: 16 weeks
Population: Full Analysis Set (participants who were randomized, received at least one dose of study treatment, and had data available for baseline and at least one post baseline evaluation). Participants who dropped out prior to Week 16, had a missing Mayo score at Week 16, or were non-responders at Week 8 are considered failures (non-remission) at Week 16.
Measure: Number; unit: Proportion of participants
Groups:
- Infliximab (IFX): IFX 5 mg/kg IV infusions administered at Weeks 0, 2, and 6 and placebo to AZA daily for 16 weeks. Responders to IFX at Week 8, will receive one more IFX infusion at Week 14; non-responders to IFX will receive placebo infusions at Weeks 8 and 10 and an additional IFX infusion at Week 14.
- Azathioprine (AZA): AZA 2.5 mg/kg orally for 14 weeks and placebo to IFX infusion at Weeks 0, 2, and 6. Responders to AZA monotherapy at Week 8 will continue on AZA therapy and receive one infliximab placebo infusion at Week 14; non-responders to AZA at Week 8 will be eligible to receive infliximab at Weeks 8, 10, and 14. This group included 20 subjects who did not respond to AZA monotherapy at Week 8 had IFX added to their treatment regimen at Weeks 8, 10, and 14.
- IFX/AZA: IFX 5 mg/kg IV at Weeks 0, 2, and 6 plus AZA 2.5 mg/kg orally daily for 16 weeks.
  Responders to IFX/AZA at Week 8 will receive one more infliximab infusion at Week 14; non-responders to IFX/AZA will receive placebo infusions at Weeks 8 and 10 and one additional infliximab infusion at Week 14.
Arm/Group | Infliximab (IFX) | Azathioprine (AZA) | IFX/AZA
Number analyzed (Participants) | 77 | 76 | 78
Proportion of participants | 0.22 | 0.24 | 0.40
Statistical Analysis 1: Comparison: Azathioprine (AZA) vs IFX/AZA; Test type: Superiority or Other; p = 0.032, Chi-squared

2. Primary Outcome: Average Remission Rate During Part 2 of the Study
Description: Due to the early termination of this study, evaluations of efficacy were not conducted for Part 2 of the study (Week 38 through Week 94 [Week 22 through Week 78 for direct entry]).
Time Frame: up to Week 94 (Week 78 for direct entry)
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Participants in Response at Weeks 8 and 16
Description: Response at Week 8 is defined as a decrease in the partial Mayo score of ≥1 point. Response at Week 16 is defined as a decrease in total Mayo score of ≥3 points and at least 30% lower than baseline Mayo score. The partial Mayo score consists of the following 3 sub-scores: stool frequency, rectal bleeding, and physician's global assessment. The total Mayo score consists of the following 4 sub-scores: stool frequency, rectal bleeding, findings of endoscopy (sigmoidoscopy), and physician's global assessment.
Time Frame: Weeks 8 and 16
Population: Full Analysis Set (participants who were randomized, received at least one dose of study treatment, and had data available for baseline and at least one post baseline evaluation). Participants who dropped out prior to Week 16, had a missing Mayo score at Week 16, or were non-responders at Week 8 are considered failures (non-responders) at Week 16.
Measure: Number; unit: Proportion of participants
Arm/Group | Infliximab (IFX) | Azathioprine (AZA) | IFX/AZA
Number analyzed (Participants) | 77 | 76 | 78
Proportion of participants
  Week 8 | 0.88 | 0.66 | 0.86
  Week 16 | 0.69 | 0.50 | 0.77

4. Secondary Outcome: Proportion of Participants With Mucosal Healing at Week 16
Description: Mucosal healing was defined as a Mayo endoscopy score of 0 or 1.
Time Frame: 16 weeks
Population: Full Analysis Set (participants who were randomized, received at least one dose of study treatment, and had data available for baseline and at least one post baseline evaluation).
Measure: Number; unit: Proportion of participants
Arm/Group | Infliximab (IFX) | Azathioprine (AZA) | IFX/AZA
Number analyzed (Participants) | 77 | 76 | 78
Proportion of participants | 0.55 | 0.37 | 0.63

5. Secondary Outcome: Proportion of Participants Who Are in Steroid-free Remission During Part 2 of the Study
Description: Due to the early termination of this study, evaluations of efficacy were not conducted for Part 2 of the study.
Time Frame: Weeks 38, 62 & 94 (Weeks 22, 46 and 78 for direct entry)
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of Participants With Mucosal Healing During Part 2 of the Study
Description: Due to the early termination of this study, evaluations of efficacy were not conducted for Part 2 of the study
Time Frame: Weeks 38, 62 and 94 (Weeks 22, 46 and 78 for direct entry)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were categorized by 3 separate timeframes: Through Week 8 (AEs reported through Week 8 of Part 1), After Week 8 (AEs reported after Week 8 through Week 16 of Part 1), and Part 2 (AEs reported during Part 2)
Groups:
- AZA Through Week 8; AZA After Week 8: Participants received AZA 2.5 mg/kg orally daily for 16 weeks. Responders to AZA monotherapy at Week 8 will continue on AZA therapy and receive one infliximab placebo infusion at Week 14; non-responders to AZA at Week 8 will be eligible to receive infliximab at Weeks 8, 10, and 14.
- IFX/AZA Through Week 8: Participants received intravenous (IV) infusions of IFX 5 mg/kg of body weight at Weeks 0, 2, and 6 plus AZA 2.5 mg/kg orally daily for 16 weeks.
  Responders to IFX/AZA at Week 8 will receive one more infliximab infusion at Week 14; nonresponders to IFX/AZA will receive placebo infusions at Weeks 8 and 10 and one additional infliximab infusion at Week 14.
- IFX Through Week 8; IFX After Week 8: Participants received IV infusions of IFX 5 mg/kg of body weight administered at Weeks 0, 2, and 6. Responders to IFX at Week 8, will receive one more IFX infusion at Week 14; non-responders to IFX will receive placebo infusions at Weeks 8 and 10 and an additional IFX infusion at Week 14.
- AZA to IFX/AZA After Week 8: Participants received AZA 2.5 mg/kg orally for 16 weeks and had IV infusions of IFX 5mg/kg of body weight added to their treatment regimen at Weeks 8, 10, and 14. Participants were either non-responders to AZA at Week 8 or had worsening of disease at Week 8.
- IFX/AZA After Week 8: Participants received IV infusions of IFX 5 mg/kg of body weight at Weeks 0, 2, and 6 plus AZA 2.5 mg/kg orally daily for 16 weeks.
  Responders to IFX/AZA at Week 8 will receive one more infliximab infusion at Week 14; nonresponders to IFX/AZA will receive placebo infusions at Weeks 8 and 10 and one additional infliximab infusion at Week 14.
- Maintenance IFX/AZA (Part 2): Participants randomized to maintenance IFX/AZA during Part 2 received IV infusion of IFX 5 mg/kg of body weight every 8 weeks (beginning at Week 22, Week 6 for direct entry) plus AZA 2.5 mg/kg of body weight daily. Four participants were from Part 1 of the study and 1 participant enrolled directly into Part 2 of the study.
- Maintenance IFX (Part 2): Participants randomized to maintenance IFX received IV infusions of IFX 5 mg/kg of body weight every 8 weeks (beginning at Week 22, Week 6 for direct entry). All participants were from Part 1 of the study.
- Intermittent IFX/AZA (Part 2): Participants randomized to intermittent IFX/AZA received IV infusions of IFX 5 mg/kg of body weight only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained) plus AZA 2.5 mg/kg of body weight daily. Three participants were from Part 1 of the study and 1 participant enrolled directly into Part 2 of the study.
- Intermittent IFX (Part 2): Participants randomized to intermittent IFX received IV infusions of IFX 5 mg/kg of body weight only upon relapse of disease (initiated at Weeks 0, 2, and 6 of individual treatment cycle and continued every 8 weeks until remission was regained). One participant from Part 1 of the study and 1 participant enrolled directly into Part 2 of the study.
- AZA (Part 2): Participants received AZA 2.5 mg/kg of body weight orally daily for Part 2 of the study. All participants were from Part 1 of the study.
- IFX/AZA (Part 2): Participants received IV infusions of IFX 5 mg/kg of body weight every 8 weeks and AZA 2.5 mg/kg of body weight orally daily until the end of the study. All participants were from Part 1 of the study.
- IFX (Part 2): Participants received IV infusions of IFX 5 mg/kg of body weight until the end of the study. All participants were from Part 1 of the study.
Arm/Group | AZA Through Week 8 | IFX/AZA Through Week 8 | IFX Through Week 8 | AZA After Week 8 | AZA to IFX/AZA After Week 8 | IFX/AZA After Week 8 | IFX After Week 8 | Maintenance IFX/AZA (Part 2) | Maintenance IFX (Part 2) | Intermittent IFX/AZA (Part 2) | Intermittent IFX (Part 2) | AZA (Part 2) | IFX/AZA (Part 2) | IFX (Part 2)
Serious Adverse Events (participants affected / at risk) | 5/79 | 4/80 | 3/78 | 0/42 | 1/20 | 0/72 | 5/74 | 0/5 | 0/2 | 0/4 | 0/2 | 1/10 | 0/48 | 3/37
Other Adverse Events (participants affected / at risk) | 27/79 | 17/80 | 17/78 | 8/42 | 3/20 | 13/72 | 9/74 | 3/5 | 1/2 | 2/4 | 0/2 | 2/10 | 12/48 | 6/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZA Through Week 8 (N=79) | IFX/AZA Through Week 8 (N=80) | IFX Through Week 8 (N=78) | AZA After Week 8 (N=42) | AZA to IFX/AZA After Week 8 (N=20) | IFX/AZA After Week 8 (N=72) | IFX After Week 8 (N=74) | Maintenance IFX/AZA (Part 2) (N=5) | Maintenance IFX (Part 2) (N=2) | Intermittent IFX/AZA (Part 2) (N=4) | Intermittent IFX (Part 2) (N=2) | AZA (Part 2) (N=10) | IFX/AZA (Part 2) (N=48) | IFX (Part 2) (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Ineffective (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileostomy closure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Anastomosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctocolectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZA Through Week 8 (N=79) | IFX/AZA Through Week 8 (N=80) | IFX Through Week 8 (N=78) | AZA After Week 8 (N=42) | AZA to IFX/AZA After Week 8 (N=20) | IFX/AZA After Week 8 (N=72) | IFX After Week 8 (N=74) | Maintenance IFX/AZA (Part 2) (N=5) | Maintenance IFX (Part 2) (N=2) | Intermittent IFX/AZA (Part 2) (N=4) | Intermittent IFX (Part 2) (N=2) | AZA (Part 2) (N=10) | IFX/AZA (Part 2) (N=48) | IFX (Part 2) (N=37)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 1 (1) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (9) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (15) | 8 (10) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Fatigue (General disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (7) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (7) | 1 (1) | 3 (4) | 0 (0) | 2 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (13) | 5 (8) | 4 (7) | 1 (1) | 0 (0) | 2 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to release and can embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to the sponsor for review. If the parties disagree on the communication, the investigator and sponsor's representative will meet for the purpose of making a good faith effort to discuss and resolve any such issues or disagreement.